CLINICAL TRIAL: NCT00517062
Title: Effects of Low Dose Growth Hormone (GH) Therapy on Insulin Sensitivity, Adipocyte Insulin-like Growth Factor-I (IGF-I) and IGF-I/Insulin Receptor Density and Regulation of Cortisol Metabolism in GH Deficient Adults
Brief Title: Low Dose Growth Hormone (GH) on Insulin Sensitivity and Cortisol Production Rates
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kevin Yuen, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB1844
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth hormone; insulin sensitivity; cortisol
MeSH Terms: conditions — Dwarfism, Pituitary; Insulin Resistance | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Growth hormone
  Interventions: Drug: Growth hormone (Genotropin)
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Growth hormone (Genotropin) — Growth hormone 0.1 mg self-injected once a day subcutaneously at bedtime.
  Other Names: Genotropin
  Arms: A
Drug: Placebo — Placebo self-injected once a day subcutaneously at bedtime.
  Other Names: Placebo.
  Arms: B

SUMMARY:
Study hypothesis:

Growth hormone (GH), through its generation of free 'bioavailable' insulin-like growth factor (IGF)-I, can improve insulin sensitivity in adults with GH deficiency.

Study aims:

The purpose of this study is to determine the mechanism of how low dose GH treatment affects the body's sensitivity to insulin actions and whether this low GH dose can affect the body's handling of steroid hormone levels (cortisol clearance) in adults with GH deficiency.

Study design:

Men and women with confirmed GH deficiency, but not recently been on GH treatment will be invited to participate in this study. The subjects will be assessed at the initial visit to ascertain their suitability before further participating in the study. If suitable, an equal number of men and women will be randomized to receive either low dose GH or placebo injection for 3 months. Before, during and after treatment, the subjects will be assessed at regularly with blood tests, scans and fat biopsies. At the first and final visit, testing will include scans to measure the amount of whole body fat and fat in the stomach area, muscle, and liver; blood tests to measure levels of cortisol, and fat tissue (taken from a biopsy) analysis to measure the density of IGF-I in the muscle; whereas blood tests to examine insulin sensitivity will also be collected. This study will use Genotropin and Genotropin pen devices, and the the data will be analyzed using a computer statistical program where the identity of the subjects will be coded to maintain confidentiality.

DETAILED DESCRIPTION:
The study will be double-blinded. One hundred subjects will be screened for eligibility initially, and 24 subjects will be enrolled with 12 subjects being randomized to receive the low GH dose (0.1 mg/day) treatment and 12 subjects to receive Placebo treatment for 3 months, allowing a 10% drop-out rate. The subjects will be taught by either by the Endocrine Nurse Specialists to self-administer the GH by subcutaneous injections using a Genotropin pen device.

Visit 1, Initial Screening Assessment (as out-patient)

* Physical examination, weight, height, and waist circumference measurements
* Fasting blood glucose levels

Visit 2, Baseline Assessment (as in-patient)

* Physical examination, weight, height, and waist circumference measurements
* Fasting blood tests for glucose, insulin, C-peptide, free IGF-I, total IGF-I, IGF-2, IGFBPs -1 and -3, non-esterified fatty acid and lipid profiles
* MRS, abdominal CT and DEXA scans
* One-step 3-hour hyperinsulinaemic euglycaemic clamp
* Cortisol production rates and urine cortisol collections
* Fat biopsies will be taken at the end of the assessment of cortisol production rates

Visit 3, Interim Assessment (Month 1) (as out-patient)

* Documentation of any adverse effects
* Fasting blood tests for glucose, insulin, C-peptide, free IGF-I, total IGF-I, IGF-2, IGFBPs -1 and -3

Visit 4, Final Assessment (Month 3) (as in-patient)

* Physical examination, weight, height, and waist circumference measurements
* Fasting blood tests for glucose, insulin, C-peptide, free IGF-I, total IGF-I, IGF-2, IGFBPs -1 and -3, non-esterified fatty acid and lipid profiles
* MRS, abdominal CT and DEXA scans
* One-step 3-hour hyperinsulinaemic euglycaemic clamp
* Cortisol production rates and urine cortisol collections
* Fat biopsies will be taken at the end of the assessment of cortisol production rates

Any extra blood remaining from the samples of blood drawn may be banked indefinitely with confidential identifiers, and may be given to researchers in the future to examine for other potential causes of diabetes and heart diseases in adults. These blood samples, however, will not be used for genetic studies.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18 to 75 years
* BMI should not exceed 40 kg/m2
* Confirmed GH deficient with at least one provocative test, e.g. insulin tolerance test and/ or GHRH/arginine
* Not received any GH therapy within last 6 months
* On a stable standardized hydrocortisone replacement dose regimen (twice a day at 8 AM and 4 PM),
* If any other pituitary hormone deficiencies are present, patient must be on optimal pituitary hormone replacement therapy, e.g. Thyroxine, testosterone and oestrogen replacement
* Normal renal and hepatic function
* Prepared to self-inject

Exclusion Criteria:

* Untreated or subclinically hypo/hyperthyroid
* Untreated or subclinically treated hypocortisolism
* Type 1 or 2 diabetes mellitus
* Subjects with evidence of nephropathy from any cause
* Subjects with evidence of retinopathy from any cause
* Any other medical illnesses that may affect the interpretation of the results
* Pregnant
* Emotional/social instability likely to prejudice study completion
* Previous history of known malignancy
* Recurrent or severe unexplained hypoglycaemia
* Known or suspected drug/alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Changes in insulin sensitivity (from the hyperinsulinemic euglycemic clamp | 3 months

SECONDARY OUTCOMES:
Changes in fat IGF-I and IGF-I/insulin hybrid receptor density and body composition. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Q. Purnell, MD, Principal Investigator — Oregon Health and Science University; Charles T. Roberts, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Yuen KC, Frystyk J, White DK, Twickler TB, Koppeschaar HP, Harris PE, Fryklund L, Murgatroyd PR, Dunger DB. Improvement in insulin sensitivity without concomitant changes in body composition and cardiovascular risk markers following fixed administration of a very low growth hormone (GH) dose in adults with severe GH deficiency. Clin Endocrinol (Oxf). 2005 Oct;63(4):428-36. doi: 10.1111/j.1365-2265.2005.02359.x. PMID 16181235
- [Background] Yuen K, Frystyk J, Umpleby M, Fryklund L, Dunger D. Changes in free rather than total insulin-like growth factor-I enhance insulin sensitivity and suppress endogenous peak growth hormone (GH) release following short-term low-dose GH administration in young healthy adults. J Clin Endocrinol Metab. 2004 Aug;89(8):3956-64. doi: 10.1210/jc.2004-0300. PMID 15292333
- [Background] Yuen K, Wareham N, Frystyk J, Hennings S, Mitchell J, Fryklund L, Dunger D. Short-term low-dose growth hormone administration in subjects with impaired glucose tolerance and the metabolic syndrome: effects on beta-cell function and post-load glucose tolerance. Eur J Endocrinol. 2004 Jul;151(1):39-45. doi: 10.1530/eje.0.1510039. PMID 15248820
- [Derived] Yuen KC, Roberts CT Jr, Frystyk J, Rooney WD, Pollaro JR, Klopfenstein BJ, Purnell JQ. Short-term, low-dose GH therapy improves insulin sensitivity without modifying cortisol metabolism and ectopic fat accumulation in adults with GH deficiency. J Clin Endocrinol Metab. 2014 Oct;99(10):E1862-9. doi: 10.1210/jc.2014-1532. Epub 2014 Jul 11. PMID 25013996
- See also: American Endocrine Society — http://www.endo-society.org/